CLINICAL TRIAL: NCT05709210
Title: Pilot Study on the Feasibility of Using Smartphone Data as a Diagnostic Marker for Alzheimer's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Collaborators: University of Poitiers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMASMART
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease; Memory Disorders
Keywords: Alzheimer Disease; Smartphone; Memory Disorders
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Memory complaint (Other)
  Interventions: Other: Recording of smartphone usage data
- Mild cognitive decline (Other)
  Interventions: Other: Recording of smartphone usage data
- Alzheimer's Disease (Other)
  Interventions: Other: Recording of smartphone usage data

INTERVENTIONS:
Other: Recording of smartphone usage data — Recording of smartphone usage data

SUMMARY:
This study will compare smartphone usage data between three groups of patients diagnosed with either a memory complaint, mild cognitive decline, or Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the leading cause of dementia in the world. The first cognitive function affected is memory and then other cognitive systems are affected leading to a progressive loss of autonomy of the patient. Currently, the diagnosis of AD is made at too late a stage. Patients with memory complaints or mild cognitive decline (MCI) are particularly at risk of developing AD.

However, there is no clinical or paraclinical evidence to predict precisely this risk of progression to AD. Investigator's hypothesis is that there is an association between the evolution of smartphone use and the conversion of cognitive status to AD.

The purpose of this pilot study is to identify existing differences between smartphone use data of patients with a memory complaint or of patients MCI or with an AD. It is a study of 90 patients (30 patients with memory complaint, 30 with MCI and 30 with AD) with a collection of smartphone usage data during three months.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting in routine care in one of the CMRR
* No sensory impairment that may compromise smartphone use

Exclusion Criteria:

* Inability to perform MMSE or MMSE < 20 ;
* Other neurodegenerative condition (Parkinson's disease, Lewy body disease, frontotemporal lobar degeneration, amyotrophic lateral sclerosis)
* Severe anxiety or depressive disorder HADS score ≥ 17
* Terminal phase of a severe disease
* Evidence of a lesion on MRI that may be involved in cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of a mathematical combination | Up to three months
  The comparison of a mathematical combination of the different parameters collected during the three months of smartphone data recording

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France